CLINICAL TRIAL: NCT05931211
Title: Translation of Motor Function to Daily Activity Performance in Individuals With SMA
Brief Title: Motor Function and Activity of Daily Life in Spinal Muscular Atrophy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202305039RINB
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-05

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will incorporate patients/ caregivers' perspectives to investigate the performance in daily activities of individuals with SMA and how it relates to their motor function abilities.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is an autosomal recessive neuromuscular disease that causes progressive muscle weakness and atrophy and eventually leads to loss of function. Despite recent advances in disease-modifying treatments, SMA can still significantly impact an individual's functioning in daily living and quality of life. This study will incorporate patients/ caregivers' perspectives to investigate the performance in daily activities of individuals with SMA and how it relates to their motor function abilities.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of SMA with genetics confirmed as 5q SMA.
* Above 3 years of age (capable of performing motor assessments).

Exclusion Criteria:

* Having severe respiratory and other medical conditions precluding safe participation in standardized motor function tests.
* Having any orthopedic surgery during the past 6 months.
* Women who are pregnant.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Spinal muscular atrophy (SMA) is an autosomal recessive neuromuscular disease that causes progressive muscle weakness and atrophy and eventually leads to loss of function.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Revised Upper Limb Module | 15-20 minutes
  The physiotherapist will perform a serious of motor test to evaluate the patient's upper limb motor function. This test is to observe the manual ability on different tasks in sitting position, including drawing along the path, opening Ziploc container, or lifting weight. And the therapist will score for each item. The Revised Upper Limb Module (RULM) are consist of 19 items. It takes about 15-20 minutes for testing.

CONTACTS AND LOCATIONS:
Overall Officials: Hsi-Wen Huang, MSc, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No